CLINICAL TRIAL: NCT06356779
Title: A National Longitudinal Study of Metastases-directed Local Ablative Therapy for Patients With Oligometastatic Disease - a Combined Interventional and Observational Trial
Brief Title: Longitudinal Study of Local Ablative Therapy in Oligometastatic Disease
Acronym: OLIGO-DK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gitte Fredberg Persson MD PhD (Other)
Responsible Party: Sponsor-Investigator, Gitte Fredberg Persson MD PhD, Associate Professor, Chief PhysicianGitte Fredberg Persson MD PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23066725
Record Dates: First submitted 2024-03-25; First posted 2024-04-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Oligometastatic Disease; Metastases; Ablation Techniques; Radiotherapy; Stereotactic Radiation; Surgery
Keywords: oligometastatic disease; metastases-directed therapy; metastasectomy; thermal ablation; stereotactic ablative radiotherapy; stereotactic radiosurgery; endpoints
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local ablative therapy (Experimental): Discussion at multidisciplinary team conferences Lesion-specific treatment plan with allocation to
  * surgical metastasectomy
  * stereotactic radiotherapy
  * thermal ablation
  * electroporation
  Interventions: Procedure: Local ablative therapy (LAT)

INTERVENTIONS:
Procedure: Local ablative therapy (LAT) — Surgical metastasectomy, stereotactic ablative radiotherapy, thermal ablation, or electroporation to all oligometastatic lesions
  Other Names: Metastases-directed therapy

SUMMARY:
This prospective national multicenter observational and interventional study aims to assess the longitudinal disease trajectory of patients with oligometastatic disease (OMD) who receive local metastasis-directed therapy. Patients with any category of OMD from any non-hematological cancer are eligible for inclusion. Local ablative therapy (LAT) includes surgical metastasectomy, radiotherapy, thermal ablation, and electroporations.

The primary objective is to assess the time to failure of LAT strategy in patients with OMD from any primary cancer treated with all LAT modalities.

DETAILED DESCRIPTION:
Patients with oligometastatic disease (OMD) are often treated with a combination of surgery, stereotactic radiotherapy, thermal ablations, or electroporation, either concurrently or in succession, however, most studies are focused on a single modality. In addition, local differences in the use of local ablative therapy (LAT) in different metastatic sites and diseases exist and may impact outcomes for patients with OMD. OLIGO-DK is designed to address these shortcomings. The aim is to offer LAT with any modality to all patients with OMD from all primary cancer histologies and in all metastatic sites, where it is deemed clinically relevant, within the framework of a national prospective multicenter study, combining both standard and non-standard LAT of OMD in an observational and an interventional cohort, respectively. At the same time, we aim to assess the longitudinal treatment trajectory of oligometastatic patients and create a national network for radiotherapy of oligometastases. Finally, we aim to create a clinically applicable prediction model for patient selection.

The trial is a national, prospective, multicentre trial. Patients with both genuine and induced non-hematological OMD who are receiving metastases-directed local ablative therapy are included, and all LAT modalities of all metastatic sites from all primary cancers are included. The trial will include both an observational cohort and an interventional cohort.

The observational cohort will include patients with OMD who are treated with LAT, which is considered standard-of-care according to national guidelines. The interventional cohort will include patients who are treated with implemented LAT techniques but for indications that are not considered standard-of-care. The final decision on treatment choice is made by the treating physician in consultation with the patient, and the patient may be referred across regional borders for specific treatments. This trial is not on its own designed for the evaluation of novel or experimental LAT techniques, where safety is a primary concern. In these cases, a separate ethical approval protocol is necessary. Patients can still be included in the OLIGO-DK protocol for prospective data collection. In addition, inclusion in this protocol does not impede patients from inclusion in other oligometastatic protocols. Patients are prospectively included, followed, and evaluated by the Centralised Trial Unit and remain included for follow-up until death or patient preference. Due to the nature of oligometastatic disease, patients may receive LAT more than once in the protocol, if the disease is amenable to further local ablative therapy.

The trial will initiate accrual in the Capital Region of Denmark, with subsequent expansion after the first interim analysis. A national OMD MDT conference and a nationwide overview of LAT options will be established during the trial. All departments of oncology, and their associated departments of surgery and interventional radiology performing LAT will be able to include patients.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology proven non-haematological cancer
* Stage IV disease
* ECOG performance status ≤ 2
* Life expectancy > 6 months
* A baseline scan within 42 days of inclusion (PET-CT or CT or MRI scan) is required, preferably within 28 days for optimal prospective evaluation
* Primary tumor must be controlled, defined by the radiographical response of the primary tumor by systemic or local treatment. If progressing, it is planned to be treated with local ablative therapy (LAT)
* Oligometastatic disease according to the ESTRO-EORTC classification, both de-novo and induced, including oligoprogression
* A maximum of five oligometastases or oligopersistent/oligoprogressive lesions. More than five metastases are allowed in the following cases, 1) location in a defined anatomical entity or 2) location in immediate proximity and as such, cannot be treated separately
* All oligometastatic lesions must be planned for definitive LAT. If all visible/progressive/persistent disease is not treated, the patient cannot be included
* Local ablative therapy must be deemed clinically relevant for the individual patient by the treating team of physicians, or a multidisciplinary team and discussion must be documented in the patient chart
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnancy
* Diffuse cancer disease, which cannot be locally ablated, i.e., leptomeningeal carcinomatosis, malignant pleural effusions, lymphangitic carcinomatosis, or peritoneal carcinomatosis
* If LAT is deemed unsafe by the MDT (e.g., tumor perforation of hollow organs)

In addition, the patients receiving SBRT to oligometastatic sites should comply with the following criteria.

* The size of the target is limited by the ability to safely deliver locally ablative doses to the metastatic lesions. Generally, an upper limit of 5 cm is recommended
* If the patient has received previous radiotherapy, the combined dose at the radiation site must not exceed the dose constraints according to Appendix 2 - Radiotherapy Recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to failure of local ablative therapy (LAT) strategy | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of LAT to progression of disease, locally or metastatically, not amenable to new LAT or progression of disease leading to initiation of or change in systemic treatment

SECONDARY OUTCOMES:
Progression-free survival | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of LAT to disease progression at any site or death
Time to widespread progression | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of LAT to disease progression not amenable to new LAT. Deaths from any cause are censored. Initiation of or change in systemic treatment is ignored
Freedom from systemic treatment | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of LAT to initiation of systemic treatment, change in systemic treatment, or end of systemic treatment due to progression. Change in or end of systemic treatment due to toxicity is ignored
Overall survival | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of first LAT to death from any cause
Time to progression | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of LAT to progression of the disease. Deaths from any cause are censored
Time to local progression | 5 years or life-long
  Defined as time from first day of LAT to progression within the treated area. In case of doubt or disagreement, the case is reviewed at the local MDT conference. Deaths from any cause are censored
Local lesion control rate at 1- and 3-years post-local ablative therapy | 3 years
  Fractions of treated lesions which have not locally progressed at 1- and 3-years after local ablative therapy. Analysed per lesion, per patient, per treatment modality and per organ
Time to distant progression | Assessed every 3-6 months for 5 years or life-long
  Defined as time from first day of LAT to progression outside the treatment field. Deaths from any cause are censored.
Investigator reported grade 3-5 CTCAE (v.5.0) LAT related toxicity | 2 years
  LAT related toxicity is defined as adverse events which are categorized by the local investigator as suspected expected or suspected unexpected due to LAT
Harms | Actively every 3-months for 2 years
  Defined as LAT-related toxicity which occurs or is worsened within 3- months of end-of-treatment (EOT). LAT-related toxicity, which occurs or is worsened after the commencement of the LAT course but before EOT, is also registered as early toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte F Persson, MD PhD, Study Chair — Copenhagen University Hospital Herlev and Gentofte; Michael RT Laursen, MD, Principal Investigator — Copenhagen University Hospital Herlev and Gentofte
Locations (11):
- Denmark (11):
  - Copenhagen University Hospital Rigshospitalet, Copenhagen, Capital Region of Denmark
  - Copenhagen University Hospital Herlev and Gentofte, Herlev, Capital Region of Denmark
  - Hillerød Hospital, Hillerød, Capital Region of Denmark
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Gødstrup Hospital, Herning, Central Jutland
  - Danish Center for Particle Therapy, Aarhus, Central Region Denmark
  - Aalborg University Hospital, Aalborg, Northern Region of Denmark
  - Zealand University Hospital, Roskilde and Næstved, Roskilde, Region Sjælland
  - Odense University Hospital, Odense, Southern Denmark Region
  - Sønderborg Hospital, Sønderborg, Southern Denmark Region
  - Vejle Hospital, Vejle, Southern Denmark Region

IPD SHARING:
Plan to Share IPD: Yes
Disease specific individual participant data will be available to the Danish Multidisciplinary Cancer Groups.
  Modality specific individual participant data will be available for separate analysis.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and the first draft of the SAP will be shared and available after the publication of the protocol article.
Access Criteria: No specific access criteria